CLINICAL TRIAL: NCT02302352
Title: Effects of Probiotics on Gastrointestinal Symptoms and on the Immune System in Patients With Systemic Sclerosis: a Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: Effects of Probiotics on Gastrointestinal Symptoms and on the Immune System in Patients With Systemic Sclerosis
Acronym: SSc
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Cristiane Kayser, MD, PhD, Associate Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/26788-3
Record Dates: First submitted 2014-11-17; First posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: Probiotics; Immune system
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Oral probiotic 1g, once/day, containing: Lactobacillus paracasei, 10x9 CFU; Lactobacillus rhamnosus,10x9 CFU; Lactobacillus acidophillus, 10x9 CFU; Bifidobacterium lactis 10x9 CFU per sachet
  Interventions: Other: Probiotic
- Placebo (Placebo Comparator): Maltodextrin 1g per sachet, once/day
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic — Probiotic 1g once a day by mouth for 8 weeks
  Other Names: Lacto Pro
  Arms: Probiotic
Other: Placebo — Maltodextrin 1g, manufactured to mimic the probiotic, once a day by mounth for 8 weeks
  Arms: Placebo

SUMMARY:
Systemic sclerosis (SSc) is an autoimmune disease with unknown etiology, which affects especially the gastrointestinal tract, lungs, heart and kidneys. Immunological abnormalities characterized by innate and acquired immune disturbances are associated with the disease development. The present study aims to evaluate the efficacy and safety of probiotics in gastrointestinal symptoms, nutritional status and innate and acquired immune responses, by means of the evaluation of IgA, Treg and Th1, Th2, and Th17 T helper subtypes levels in patients with SSc. In addition the levels of CD4+ T helper Th1, Th2 and Th17 subtypes and Treg levels will be compared to a healthy control group.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a chronic autoimmune disease, which affects the gastrointestinal tract, lungs, heart and kidneys. A shift in the balance between T helper 1 (Th1) and Th2 subtypes and between regulatory T cells (Treg) and Th17 cells levels, as well as intestinal microbiota abnormalities may be present in SSc. These abnormalities can stimulate inflammatory response, and cause intestinal epithelial damage. The use of oral probiotics for microbiome or immune response modulation can be attractive especially in autoimmune diseases. Objectives: To evaluate the efficacy and safety of probiotics in gastrointestinal symptoms, nutritional status and innate and acquired immune responses, by means of the evaluation of IgA, Treg and Th1, Th2, and Th17 T helper subtypes levels in patients with SSc. In addition the levels of CD4+ T helper Th1, Th2 and Th17 subtypes and Treg levels will be compared to a healthy control group. Patients and methods: A randomized double-blind placebo-controlled clinical trial, with 76 SSc patients will be performed. Patients will be randomly assigned to receive oral probiotics once a day or placebo for 8 weeks. The primary outcome will be changes in the gastrointestinal symptoms between baseline and week 8. Clinical evaluation, scleroderma Health Assessment Questionnaire (sHAQ), food intake record, anthropometry assessment and laboratory evaluation will be performed at baseline (T0), at week 4 (T1) and week 8 (T2). C-reactive protein (CRP) and immunoglobulin A (IgA) serum levels assessment will be performed at each visit. The proportion of CD4+ and CD8+ T cells, and Tregs (CD4+CD25+Foxp3+CD127low), and Th1, Th2 e Th17 CD4+ T cell subsets levels will be evaluated using flow cytometer at each visit in SSc patients and also in 50 healthy subjetcs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic sclerosis according to the 2013 ACR/EULAR classification criteria for SSc;
* Patients with gastrointestinal symptoms related to SSc including: gastrointestinal reflux, bloating, diarrhea and constipation;
* Written informed consent provided by the subjects.

Exclusion Criteria:

* Overlap syndromes with systemic lupus erythematosus, polymyositis/dermatomyositis and rheumatoid arthritis;
* Use of antibiotics and/or probiotics four weeks before baseline;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-04 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the gastrointestinal symptoms as measured by the "The University of California Los Angeles Scleroderma Clinical Trials Consortium Gastrointestinal Tract 2.0 (GIT 2.0)" Questionnaire | baseline and eight weeks

SECONDARY OUTCOMES:
Scleroderma Health Assessment Questionnaire (sHAQ) | baseline and eight weeks
Food intake record | baseline and eight weeks
Anthropometry assessment as measured by the body mass index (BMI) | baseline and eight weeks
C-reactive protein (CRP) and immunoglobulin A (IgA) serum levels | baseline and eight weeks
Proportion of CD4+ and CD8+ T cells | baseline and eight weeks
Tregs (CD4+CD25+Foxp3+CD127low) levels | baseline and eight weeks
Th1, Th2 and Th17 CD4+ T cell subsets levels | baseline and eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Kayser, Principal Investigator — Associate Professor
Locations (1):
- Systemic Sclerosis Outpatient Clinic, Hospital São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Marighela TF, Arismendi MI, Marvulle V, Brunialti MKC, Salomao R, Kayser C. Effect of probiotics on gastrointestinal symptoms and immune parameters in systemic sclerosis: a randomized placebo-controlled trial. Rheumatology (Oxford). 2019 Nov 1;58(11):1985-1990. doi: 10.1093/rheumatology/kez160. PMID 31056685